CLINICAL TRIAL: NCT02454374
Title: Joint Loading vs Normal Physiotherapy Care in Degenerative Knees (V1)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leeds Comunity Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP0159
Record Dates: First submitted 2015-04-15; First posted 2015-05-27 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Osteo Arthritis Knee
Keywords: Physiotherapy; Knee Loading; Randomised Controlled Trial; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Knee Loading (Experimental): Progressive joint loading intervention will be taught by a program of exercises by the treating physiotherapist. The intervention consists of knee flexion (bending) and knee extension (straightening). Participants will be assessed for their immediate response to treatment during each assessment or treatment session and advised on the appropriate level of self-directed exercises to be performed twice daily. The clinician will review the patient at follow up appointments during the treatment period, progressing to the next level of exercises or by increasing intensity, duration or repetitions as appropriate. The physiotherapist will encourage compliance during the treatment period and beyond
  Interventions: Procedure: Knee Loading protocol
- Routine physiotherapy care (Active Comparator): Normal care delivered to the control group will be based on current NICE guidelines (2014) for non-pharmacological management of OA which includes verbal and written advice/education; education regarding weight loss; exercise to include local muscle strengthening and general aerobic fitness; with or without manual therapy. Clinicians will be asked to refrain from using the progression of techniques specifically documented in the progressive loading protocol (not currently considered to constitute 'normal care'). Treating clinicians will be asked to record specific exercises and manual therapy techniques employed in the patient's records. Participants will be asked to complete a home treatment record sheet.
  Interventions: Procedure: Routine Physiotherapy Care

INTERVENTIONS:
Procedure: Knee Loading protocol — The clinician will review the patient at follow up appointments a further two to four times during the treatment period (dependent on symptom resolution/response), progressing to the next level of exercises or by increasing intensity, duration or repetitions as appropriate (each participant will be asked to maintain a home treatment diary sheet). The physiotherapist will encourage compliance during the treatment period and beyond.
  Arms: Knee Loading
Procedure: Routine Physiotherapy Care — Routine Physiotherapy Care
  Arms: Routine physiotherapy care

SUMMARY:
This study is a randomised controlled clinical trial designed to evaluate the effectiveness of two different exercise based treatments in the management of patients with knee problems related to degenerative (wear and tear) changes.

Recent evidence suggests that putting weight through a joint (joint loading) may be beneficial.

The Investigators know that physiotherapy and exercise is important in treating these patients, but the investigators do not know which exercises work best. In this study the investigators will be comparing current physiotherapy care against a new programme of exercises that gradually increases the amount of joint loading.

The study will recruit approximately 140 patients from the Leeds Musculoskeletal (MSK) service, who are over the age of 45 and have been referred for physiotherapy by their GP for activity related knee pain.Patients who are suitable and happy to take part will be selected randomly (not chosen by the patient or physiotherapist) to receive either normal physiotherapy treatment, or the knee loading exercises. The treatment phase will last for six weeks and participants will be asked to carry out their exercises twice daily during this time. At the end of this period, patients will be asked tocomplete questionnaires and again at six months so that the investigators can assess how the patients are doing.

The main aim is to evaluate clinical effectiveness of the progressive joint loading protocol. However, the data collected will also be used to see if there is a way of identifying in advance those who might respond better to either treatment.

The investigators will also collect some information relating to the cost effectiveness of delivering different treatments. The final aim of this study is to test how easy it is to collect more detailed data in this area if a related study were to be carried out in the future.

DETAILED DESCRIPTION:
The Leeds University academic partner will provide statistical support for the study team during the data analysis phase. Predictor variables with a substantial single variable association with each outcome (p<0.2) will be included in a multivariable linear regression model to determine the adjusted associations of improved outcome from being in the treatment arm. A second model will use multi-levels (two levels: 1. time points for individuals, 2. individuals) to determine whether the trajectory of change in outcome scores differs between the two arms of the study. Significant predictors of improved outcomes will be determined from both of these models. A sensitivity analysis will be undertaken for final models based on degrees of compliance to home treatment using categories determined through exploratory analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred to the Leeds Community Healthcare Musculoskeletal service aged 45 years or over with primary symptoms suggestive of degenerative intraarticular knee pain with a dominant mechanical presentation (i.e. activity related pain, functional limitation, morning stiffness not exceeding 30 minutes) AND
2. Limitation in weightbearing range of motion of the knee joint (tibiofemoral joint limitation in flexion or extension)

Exclusion Criteria:

1. Subjects with cognitive impairment or medical conditions preventing understanding or participation in the study
2. Subjects with symptoms requiring surgical evaluation or other intervention
3. Knee symptoms related to pathology other than degenerative intraarticular pathology
4. Subjects who are contraindicated from kneeling or crouching
5. Subjects unable to attend the full study programme

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome score (KOOS) | 6 and 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven Foster, Principal Investigator — Leeds Community Healthcare NHS Trust
Locations (1):
- Leeds Musculosktal Servive, Leeds, United Kingdom